CLINICAL TRIAL: NCT00322634
Title: Investigator Initiated Trial: Prospective Study of Clinical Predictors of Survival in Cancer Patients With Metastatic Solid Tumors
Brief Title: Clinical Predictors of Survival in Cancer Patients With Metastatic Solid Tumors
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0535C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2011-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The use of performance status and LDH in combination can predict patient survival more accurately than physician clinical impression or the patients' own feelings about their survival

DETAILED DESCRIPTION:
Patients with incurable cancer frequently ask their doctors for an estimate of survival. Such estimates can assist patients in making decisions about how best to spend their time and energy. Survival estimates are also required when considering patients with incurable cancer for experimental treatments. However, such estimates are difficult to make. There is some data to suggest that a simple clinical measure, the performance status, combined with a laboratory blood test, the LDH, may assist in making the survival estimate more realistic. This study is designed to test if this is the case, using patients with metastatic lung, breast, colorectal, prostate, or pancreatic cancer or patients with cancer of unknown primary who have exhausted life-prolonging therapy. These patients will be asked to consent to entering this study. Their performance status will be assessed by the Karnofsky and WHO scales, they will be asked to have their blood tested for LDH and they and their doctor will be asked to estimate their survival. After study entry they will be allowed to receive palliative radiotherapy, surgery or systemic therapy as indicated including protocol treatment. After study entry, the only other requirement is that the date of the patients death be reported so that the duration of survival can be compared with the doctors and patients estimate and correlated with the performance status and LDH.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be at least 18 years of age
2. All patients must have documented incurable metastatic cancer
3. All patients must have exhausted any treatments which are known to prolong survival in their disease, or have elected not to receive further life-prolonging therapy. Specifically, patients with the following are eligible:

   1. Non-small cell lung cancer patients after third systemic therapy
   2. Small cell lung cancer patients after second systemic therapy
   3. Breast cancer patients after third cytotoxic therapy (does not include hormonal therapy)
   4. Colorectal cancer patients after second systemic therapy
   5. Hormone refractory prostate cancer patients after first cytotoxic therapy
   6. Cancer of unknown primary
   7. Pancreatic cancer patients after first systemic therapy
4. The use of systemic (chemotherapy, immunotherapy) or local treatments (XRT) for palliation of symptoms is allowed
5. Patients with a history of previous cancers are allowed
6. Patients with a history of other significant disease (e.g. heart disease, COPD, etc.) are allowed
7. All patients must sign informed consent

Exclusion Criteria:

1. Patients with acute or chronic leukemia, Hodgkin's disease, or non-Hodgkins lymphoma are excluded
2. Patients who do not sign informed consent are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic solid tumors.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Disease Progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Purdy, MD, Principal Investigator — Hematology & Oncology Associates
Locations (5):
- United States (5):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Radiation Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - St. Vincent Regional Medical Center, Santa Fe, New Mexico